CLINICAL TRIAL: NCT06073223
Title: Pilot Study of an Intervention to Decrease Overtreatment of Patients With Low-risk Thyroid Cancer
Brief Title: Intervention to Decrease Overtreatment of Patients With Low-risk Thyroid Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UMCC 2023.009; HUM00218043 (Other: University of Michigan); R03CA283105 (NIH)
Record Dates: First submitted 2023-09-26; First posted 2023-10-10 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Who Masked: Participant
Masking Description: The control group will be blinded to the intervention and receive usual care, which involves providing no disease or treatment specific information outside the surgeon visit.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CQUPLE Intervention (Experimental): A novel intervention called CQUPLE (pronounced "couple"), which includes two interventions delivered together: (1) a Chart of side-by-side, evidence-based information comparing all three treatment options for low-risk thyroid cancer, including expected outcomes and (2) a Question Prompt List that contains key questions to consider asking the surgeon.
  Interventions: Other: CQUPLE
- Usual Care Control (Active Comparator): The control group will receive usual care, which involves providing no disease or treatment specific information outside the surgeon visit.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Usual Care — The control group will receive usual care, which involves providing no disease or treatment specific information outside the surgeon visit.
  Arms: Usual Care Control
Other: CQUPLE — Our research team developed a novel intervention called CQUPLE (pronounced "couple"), which includes two interventions delivered together: (1) a Chart of side-by-side, evidence-based information comparing all three treatment options for low-risk thyroid cancer, including expected outcomes and (2) a Question Prompt List that contains key questions to consider asking the surgeon. The intervention is grounded in social cognitive theory and aims to increase patient awareness of treatment options and their outcomes, patient activation, and self-efficacy for decision making.
  Arms: CQUPLE Intervention

SUMMARY:
The study will include 50 patients newly diagnosed with low-risk thyroid cancer ranging from 18-80 years of age. After scheduling their surgeon visit, the investigators will enroll patients and measure their intended treatment choice, baseline awareness of the three treatment options, expected outcomes, self-efficacy, and activation. The participants will then be randomized 1:1 and deliver the CQUPLE intervention to the intervention group. The control group will receive usual care, which involves providing no disease or treatment specific information outside the surgeon visit. The study team will repeat all measures prior to the surgical consult and after the surgical consult. The study team will record the patients' actual treatment choice after the consult.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 80 years
* Low risk papillary thyroid cancer or highly suspicious for cancer

  * Low risk papillary thyroid cancer

    * cT1-2: Tumor size 4 cm or smaller and limited to the thyroid on ultrasound
    * cN0: No evidence of lymph node metastasis on ultrasound
    * cM0: No evidence of distant metastasis on imaging
  * Highly suspicious for cancer

    * Cytology meeting Bethesda V or Bethesday III or IV with molecular testing indicating a 70% risk of greater of thyroid cancer
    * Nodule size 4 cm and smaller
    * Limited to the thyroid on ultrasound
    * No evidence of suspicious lymph nodes
    * No evidence of thyroid cancer outside of the neck
* Referred for surgical consultation.

Exclusion Criteria:

* History of previous thyroid cancer or thyroid surgery and parathyroid surgery
* Non-English speaking
* Deaf

Subject Selection (for Surgeons)

Surgeon Inclusion Criteria

* Performs at least one thyroid surgery annually on adults
* Credentialed at Michigan Medicine

Surgeon Exclusion Criteria

* None

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-09-18 (Actual); Primary Completion 2025-12-20 (Actual); Study Completion 2025-12-20 (Actual)

PRIMARY OUTCOMES:
Acceptability of the CQUPLE intervention to patients | day after clinic visit
  This 4-item quantitative instrument assesses participants' views on the acceptability of a novel intervention, such as CQUPLE. The response option are on a 5-point scale from 'completely disagree' to 'completely agree.' Scales are created for each measure by averaging responses. Scale values range from 1 to 5. No items need to be reverse coded. Interventional group only.
Acceptability of the CQUPLE intervention to providers | at time of surgery
  This 15-question quantitative instrument measures physician acceptability of decision support interventions with respect to ease of use and approach. Response options are on a 5-point Likert scale from 1 to 5 ('strongly disagree' to 'strongly agree'). Responses are reported descriptively in terms of proportions responding positively or negatively on each criterion.
Feasibility of the CQUPLE intervention (recruitment) | up to 7 days after surgery
  Recruitment rate will be defined as the number of patients who confirm eligibility during the screening process (they can be screened by phone or by questions in Qualtrics prior to consent) divided by the number who consent to participate.
Feasibility of the CQUPLE intervention (retention) | up to 7 days after surgery
  Retention will be defined as the number who complete the entire study (pre- and post-assessments) divided by the number consented.
Feasibility of the CQUPLE intervention (burden of data collection on study team) | up to 7 days after surgery
  To measure burden of data collection, the investigators will record the number of emails, texts, and phone calls needed for each participant to complete the measures.

SECONDARY OUTCOMES:
Effect of CQUPLE on patient treatment choice | baseline, pre-visit and post visit- up to 7 days
  The investigators will assess patient's intended treatment choice at baseline and pre-visit. The investigators will assess actual treatment choice post-visit. The investigators will ask: "Knowing what you know now, which treatment option would/did you choose for yourself?" Answers will include: removal of the entire thyroid, removal of half of the thyroid, surveillance with ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Pitt, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- The University of Michigan Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will make de-identified data available on a by request basis and will require a DUA
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: A data set comprised of survey data, interview and conversation transcripts, and metadata will be made available for non-profit research purposes within one year of the completion of the funded project period or upon acceptance of the data for publication, whichever is earlier.
Access Criteria: The data set will be made available to external investigators and the public on a case-by-case basis, to be approved by the PI and in accordance with institutional, HIPAA, state and federal regulations. A data-sharing agreement may be instituted, depending upon the data to be shared.